CLINICAL TRIAL: NCT04384731
Title: Randomized Controlled Phase II Trial of Poractant Alfa (Curosurf®) by Fiberoptic Bronchoscopy-directed Endobronchial Administration in Acute Respiratory Distress Syndrome (ARDS) Due to COVID-19 Viral Pneumonia
Brief Title: Curosurf® in Adult Acute Respiratory Distress Syndrome Due to COVID-19
Acronym: Caards-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Christophe LENCLUD (Other)
Responsible Party: Sponsor-Investigator, Dr Christophe LENCLUD, Principal Investigator, Versailles Hospital
Organization: Versailles Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20/06
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: COVID-19; ARDS, Human
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — poractant alfa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surfactant arm (Experimental): patient receiving the surfactant
  Interventions: Drug: poractant alfa
- Control arm (No Intervention): patient not receiving the surfactant

INTERVENTIONS:
Drug: poractant alfa — Patient receiving surfactant (3 mL/kg of a poractant alpha solution diluted to 16 mg/mL, resulting in a total dose of 48mg/kg) administred by bronchial fibroscopy. The total volume will be divided in each of the five lobar bronchi.
  Arms: Surfactant arm

SUMMARY:
Surfactant replacement therapy (SRT) improves oxygenation and survival in NRDS and some infant ARDS. SRT was tried in adult ARDS with conflicting results. Research by Filoche and Grotberg helped to understand the failure of previous clinical trials and yielded a strong scientific rationale for SRT success, now allowing to design a new administration protocol for SRT in adults, to be tested by this clinical trial in COVID-19 adult ARDS patients.

Patients will be randomized to receive either a bronchial fibroscopy alone (with aspiration of secretions) or a bronchial fibroscopy with administration of 3 mL/kg of a solution of poractant alpha diluted to 16 mg/mL and distributed into each of the 5 lobar bronchi.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years
* Intensive care unit admission.
* Intubation and mechanical ventilation since less than 72h.
* Positive end-expiratory pressure ≥ 5 cmH2O.
* Acute respiratory distress syndrome following Berlin definition.
* COVID-19
* PaO2/FiO2 ratio < 150 mmHg during at least 3 hours despite PEP trial.
* Compliance of the respiratory system < 50 mL/cmH2O

Exclusion Criteria:

* Contraindication to prone position.
* Pregnancy.
* Weight < 40 kg
* height < 140 cm or height > 190 cm.
* Profuse bronchorrhea (at least 1 succion per hour during 3 hours).
* Other significant cause than ARDS to the respiratory failure.
* Decision to limit active therapies.
* No arterial line in place.
* Obesity with weight / height ratio > 1 kg / cm.
* Impossible to give neuromuscular blockers (e.g. drug unavailable owing to global pandemia).
* Severe chronic respiratory failure with oxygen at home.
* Other severe acute or chronic organ faillure (eg severe liver cirrhosis, severe chronic cardiac failure).
* History of pneumonectomy or pulmonary lobectomy.
* Patient scheduled for extracorporeal membrane oxygenation.
* Known hypersensibility to Curosurf.
* Contraindication to bronchial fibroscopy.
* Person under legal protection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-05-29 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of the PaO2 / FiO2 ratio between the measurements taken before (t0) and one hour after the end of the invasive procedure (H1). | 1 hour post treatment

SECONDARY OUTCOMES:
Oxygenation : PaO2 / FiO2 ratio. | up to Day 1 and up to Day 7
Oxygenation : area under the PaO2 / FiO2 curve. | up to Day 1 and up to Day 7
Oxygenation : area under the SpO2 curve. | up to Hour 1 and up to Hour 24
Evolution of thoraco-pulmonary compliance (mL / mbar) between before and one hour after the procedure. | 1 hour
Overall survival rate | at 28 days, 56 days.
Mortality rate at discharge from the intensive care unit. | through study completion, an average of 6 months.
Mortality rate at discharge from the hospital. | through study completion, an average of 6 months.
Number of ventilator-free days | Day 28, Day 56
Number of prone position sessions. | up to 56 days
Time between inclusion and the last prone position session. | up to 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LENCLUD, MD, Principal Investigator — Hospital of Mantes-la-Jolie, France
Locations (1):
- CH Francois Quesnay, Mantes-la-Jolie, France

IPD SHARING:
Plan to Share IPD: No